CLINICAL TRIAL: NCT04006938
Title: The Effect of Continuous Versus Intermittent Aerobic Exercise on Glycemic Control in a Barbadian Population With Type 2 Diabetes - A Crossover Randomized Control Trial
Brief Title: Effect of Continuous vs Intermittent Aerobic Exercise on Glycemic Control in a Barbadian Population With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Springfield College (Other)
Responsible Party: Principal Investigator, Kristyn Kirton, Principal Investigator, Springfield College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KCK00000001
Record Dates: First submitted 2019-06-29; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The proposed study is a crossover randomized controlled study. There will be two intervention groups - a single 30-minute bout of moderate intensity aerobic exercise before breakfast and three (3) 10-minute bouts of moderate intensity aerobic activity before breakfast, lunch and dinner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Bout ('S') - 30 minutes of moderate intensity cycling (Experimental): Subjects will perform a single 30-minute bout of moderate intensity cycling before breakfast
  Interventions: Behavioral: Single Bout ('S')
- Multiple Bout ('M') (Experimental): Subjects will perform three (3) 10-minute bouts of moderate intensity cycling before breakfast, lunch and dinner
  Interventions: Behavioral: Multiple Bout ('M')

INTERVENTIONS:
Behavioral: Single Bout ('S') — Each subject will perform a single bout of 30-minutes of moderate-intensity cycling before breakfast
  Arms: Single Bout ('S') - 30 minutes of moderate intensity cycling
Behavioral: Multiple Bout ('M') — Each subject will perform three (3) 10-minute bouts of moderate intensity cycling before breakfast, lunch and dinner
  Arms: Multiple Bout ('M')

SUMMARY:
The purpose of this study will be to evaluate and compare the effect of a single 30-minute bout of moderate intensity aerobic exercise to the effect of three 10-minute pre-prandial bouts of energy-matched and volume-matched aerobic exercise on 2-hr post prandial and fasting blood sugar levels, in a sample of type 2 diabetes patients, aged 30-65 years, living in Barbados

Research Hypotheses:

The three bouts of pre-prandial moderate intensity aerobic exercise will result in lower post prandial blood sugar levels when compared to the single bout of moderate intensity aerobic exercise.

The three bouts of pre-prandial moderate intensity aerobic exercise will result in lower fasting blood sugar levels on the morning following the exercise intervention when compared to the single bout of moderate intensity aerobic exercise

DETAILED DESCRIPTION:
With the background that there is increasing evidence that breaking up sedentary time with physical activity may be potentially associated with improved blood glucose levels (Francois et al., (2014) & van Dijk et al., (2013), this study aims to investigate and compare the effect of a single 30-minute bout of moderate intensity aerobic exercise to the effect of three 10-minute pre-prandial bouts of energy-matched and volume-matched aerobic exercise on 2-hr post prandial and fasting blood sugar levels in a sample of type 2 diabetes patients.

Different from previous studies, this research seeks to evaluate these effects in a Black Caribbean population, in a type 2 diabetes population on medication including insulin and also seeks to evaluate if either exercise regimen is indeed palatable to the target population by evaluating treatment acceptability.

The proposed study will be a crossover randomized controlled study. There will be two intervention groups - a single 30-minute bout of moderate intensity aerobic exercise before breakfast and three (3) 10-minute bouts of moderate intensity aerobic activity before breakfast, lunch and dinner. The primary outcome measure will be 2-hr post prandial blood sugar levels and fasting blood sugar levels on the day following the intervention. Neither subject nor investigator will be blinded to the intervention.

Subjects will include patients with a documented diagnosis of type 2 diabetes, that is a documented HbA1C ≥ 6.5%. Baseline data will include body mass and body composition and will be measured using the bioelectrical impedance technique (Tanita scale). Waist circumference will be assessed using a Gulick tape measure. Baseline sedentary behaviour and physical activity level will be assessed using the validated International Physical Activity Questionnaire.

All recruited subjects will be asked to complete two exercise interventions separated by a one-week washout period: 1) a single 30-minute bout of moderate intensity aerobic exercise before breakfast and 2) three (3) 10-minute bouts of moderate intensity aerobic activity before breakfast, lunch and dinner. Each subject will be randomized to one of two treatment sequences: single bout followed by multiple bouts (S-M) or multiple bouts followed by single bout (M-S). The randomization will be done using online statistical computing web programming (www.randomization.com) to generate a randomization schedule with balanced permutations.

Timing between exercise completion and commencement of meal intake will be approximately 15 minutes. A heart rate reserve range of 40-59% will be used to define moderate intensity. Heart rate will be measured using a validated Polar heart rate monitor. Rate of perceived exertion will be a secondary measure of exercise intensity.

Two-hour (2hr) post prandial blood sugar levels and fasting blood sugar levels on the day following the exercise intervention will be measured using a validated capillary blood glucose meter. Blood pressure will also be measured at the same times that blood glucose values are taken using a validated automated blood pressure machine.

Standardized meals of fixed nutrient content and individualized to the subject's calculated estimated daily caloric requirements will be provided to subjects on the day of the exercise interventions. Treatment acceptability will be assessed following each exercise intervention using an expert-designed questionnaire that will be piloted in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-65 years
* Documented diagnosis of type 2 diabetes (HbA1C ≥ 6.5%)

Exclusion Criteria:

* Subjects currently managed on prandial insulin
* Subjects who have recently started insulin (within the previous month)
* Subjects with a history of frequent hypoglycemic episodes within the previous 2 weeks,
* Pregnancy
* Subjects with a history of cerebrovascular accident, myocardial infarction, chronic kidney disease, autonomic and peripheral neuropathy
* Subjects with contraindications to exercise according to ACSM 2018 guidelines

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
2 hour post prandial blood glucose level after breakfast | single point measurement taken 2 hours after breakfast consumption
  blood glucose level 2 hours after breakfast consumption
2 hour post prandial blood glucose level after lunch | single point measurement taken 2 hours after lunch consumption
  blood glucose level 2 hours after lunch consumption
2 hour post prandial blood glucose level after dinner | single point measurement taken 2 hours after dinner consumption
  blood glucose level 2 hours after dinner consumption
Fasting blood sugar level | single point measurement taken after 8 hours of fasting
  blood sugar level after 8 hours of fasting performed on day following exercise intervention

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Headley, PhD, Study Chair — Springfield College

REFERENCES:
- [Background] Francois ME, Baldi JC, Manning PJ, Lucas SJ, Hawley JA, Williams MJ, Cotter JD. 'Exercise snacks' before meals: a novel strategy to improve glycaemic control in individuals with insulin resistance. Diabetologia. 2014 Jul;57(7):1437-45. doi: 10.1007/s00125-014-3244-6. Epub 2014 May 10. PMID 24817675
- [Background] van Dijk JW, Venema M, van Mechelen W, Stehouwer CD, Hartgens F, van Loon LJ. Effect of moderate-intensity exercise versus activities of daily living on 24-hour blood glucose homeostasis in male patients with type 2 diabetes. Diabetes Care. 2013 Nov;36(11):3448-53. doi: 10.2337/dc12-2620. Epub 2013 Sep 16. PMID 24041682
- [Background] American College of Sports Medicine. (2018). ACSM's guidelines for exercise testing and prescription (5th edn.). Philadelphia, PA: Lippincott Williams & Wilkins.